CLINICAL TRIAL: NCT07241208
Title: Effect of Combined Use of Flexible Bronchoscope on First-attempt Sucess in Tracheal Double Lumen Tube Intubation Using Videolaryngosocpe: A Randomized Controlled Trial
Brief Title: Comparison of Double-lumen Tube Intubation Between Fiberoptic Bronchoscopy and Video Laryngoscope
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Hyungseok Seo, MD, PhD, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC_IRB_202508009001
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: One Lung Ventilation in Thoracic Surgery
Keywords: double-lumen tube; one lung ventilation; video laryngoscopy; flexibe bronchoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VL (No Intervention): DLT intubation using video laryngoscope only
- VL+FOB (Active Comparator): DLT intubation using video laryngoscope and fiberoptic bronchoscope
  Interventions: Procedure: Fibertoptic Bronchoscopy

INTERVENTIONS:
Procedure: Fibertoptic Bronchoscopy — Use Fibertopic bronchoscopy for DLT intubation
  Arms: VL+FOB

SUMMARY:
The goal of this clinical trial is to compare the first-attempt success rate in double-lumen tube intubation. The main question it aims to answer:

Is there any difference in the first-attempt success rate of intubation between using flexible bronchoscopy and a video laryngoscope? Researchers will compare the group using a flexible bronchoscope and video laryngoscope with the group using a video laryngoscope only to see if there is a difference in first-attempt success rate.

Participants will be intubated in one of two interventions.

DETAILED DESCRIPTION:
For double-lumen tube insertion, a video laryngoscope can usually be used. However, because the camera is located at the tip, there can be a difference between the line of sight and the actual glottic view, which may make double-lumen tube steering difficult.

Flexible bronchoscopy can guide the double-tube along the natural curvature of the airway with less trauma. In the present research, we hypothesized that the first-pass success rate may differ between a group using video laryngoscopy only and a group using video laryngoscopy and flexible bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled operation
2. Patients required to double lumen tube insertion for thoracic surgery
3. ASA PS 1, 2, 3

Exclusion Criteria:

1. BMI <18.5 or 35.0
2. history of airway surgery
3. suspicious of high aspiration risk
4. Pathology in oropharynx or larynx such as tumor, poly, or inflammation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
first attempt success rate | from enrollment to the end of tracheal intubation
  The proportion of successful intubation at the first attempt

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
There can be a national policy for securing individual participant data